CLINICAL TRIAL: NCT04348513
Title: Triiodothyronine for the Treatment of Critically Ill Patients With COVID-19 Infection (Thy-Support)
Brief Title: Triiodothyronine for the Treatment of Critically Ill Patients With COVID-19 Infection
Acronym: Thy-Support
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to specific inclusion criteria no more subjects could be enrolled.
Sponsor: Uni-Pharma Kleon Tsetis Pharmaceutical Laboratories S.A. (Industry)
Collaborators: Attikon Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: T3inj-02/ThySupport
Record Dates: First submitted 2020-04-09; First posted 2020-04-16 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Pulmonary Infection; Covid-19
Keywords: Covid-19; Pulmonary Infection; T3; Triiodothyronine; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Phase II, parallel, prospective, randomized, double-blind, placebo controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T3 solution for injection (Experimental): T3 Solution for injection 10 μg/ml, each vial contains 150μg of liothyronine in a total volume of 15ml. The dose administered will be 0.8g/kg i.v. bolus starting within 60min after respiratory support and will be followed by an infusion of 0.113g. kg-1.h-1 i.v. for 48 hours (therapeutic dose). After the first 48h, a maintenance dose will be administered corresponding to 50% of the therapeutic dose (0.057g. kg-1.h-1 i.v.). Drug administration will stop after successful weaning or end of followup (maximum 30 days).
  Interventions: Drug: T3 solution for injection
- Placebo (Placebo Comparator): Composition identical apart from the active substance. Same dosage.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: T3 solution for injection — For example, for a patient of 77Kg of weight, a dose of 6ml (60 μg) will be administered as a bolus intravenously over 2-3 min within 60 min of respiratory support initiation. Then, the patient for the next 24 hours will receive 21ml of the product (total of 210 μg of T3) that will be diluted in NaCl 0.9% and administered with a pump at a steady flow rate of 10.4 ml/h for a total duration of 48 hours. From day 3 till successful weaning or end of follow-up, the patient will receive 50% of this dose, 10.5 ml of the product (total of 105 μg of T3) that will be diluted in NaCl 0.9% and administered with a pump at a steady flow rate of 5.2 ml/h.
  Arms: T3 solution for injection
Drug: Placebo — Same as with T3 solution for injection.
  Arms: Placebo

SUMMARY:
This study is a phase II, parallel, prospective, randomized, double-blind, placebo controlled trial. The present study will aim to address the efficacy and safety of acute administration of triiodothyronine on ICU patients diagnosed with pulmonary infection due to COVID-19 and require mechanical respiratory support or ECMO.

DETAILED DESCRIPTION:
It seems that thyroid hormone is critical in the response to body injury and is now considered as potential pharmaceutical intervention to limit acute tissue injury. TH (via its regulation of stress induced p38 MAPK activation) exerts antiapoptotic action and protects tissue from injury, with additional favorable effects on immune system and on viral load in infected tissue. This may be a novel and more effective treatment for critically ill viral infected patients.

ThyRepair is the first study which is underway and investigates the safety and efficacy of high dose T3 treatment in patients with acute myocardial infarction undergoing primary angioplasty. The preliminary reports show that this treatment is safe and the efficacy on tissue repair is promising. This therapeutic modality could also be tested in the acute setting of sepsis in which thyroid hormone is involved in the pathophysiology of multi-organ dysfunction. The safety and efficacy of T3 on heamodynamics in sepsis has been previously demonstrated in a small trial.

The present study is phase II, parallel, prospective, randomized, double-blind, placebo controlled trial which aims to investigate the potential effect of T3 intravenous use in the recovery of critically ill patients admitted in ICU due to COVID19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with pulmonary infection due to COVID-19, admitted in ICU and require mechanical ventilation or ECMO
* Male and female with Age>18 years old
* Signed informed consent from patient or relatives

Exclusion Criteria:

* Pregnant or breast-feeding women
* Severe systemic disease (cancer, auto-immune etc) before infection accompanied by reduced life expectancy <6 months
* Participation in another trial of an investigational drug or device
* Corticosteroid Use before initiation of treatment
* Sympathomimetic Use before initiation of treatment (epinephrine, norepinephrine, dobutamine, dopamine, phenylephrine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Assessment of weaning from cardiorespiratory support | 30 days
  The primary objective of the study is to determine whether the administration of intravenous triiodothyronine in ICU patients diagnosed with pulmonary infection due to COVID-19 facilitates weaning from cardiorespiratory support compared to placebo. Successful weaning is defined as no requirement for ventilatory support after extubation (mechanical support) or support from ECMO for 48 hours. The primary objective will be measured as percentage of patients successfully weaned after 30 days of follow-up.

SECONDARY OUTCOMES:
Assessment of hemodynamic status | 30 days
  Hemodynamic status will be assessed by continuous blood pressure measurements (systolic BP in mmHg)
Assessment of hemodynamic status | 30 days
  Hemodynamic status will be assessed by continuous blood pressure measurements (diastolic BP in mmHg)
Assessment of hemodynamic status | 30 days
  Hemodynamic status will be assessed by continuous blood pressure measurements (mean BP in mmHg)
Assessment of hemodynamic status | 30 days
  Hemodynamic status will be assessed by the number of participants with use of inotropic and vasoactive drugs
Assessment of pulmonary function | 30 days
  Pulmonary function will be assessed by arterial measurement of blood gases (arterial partial pressure of oxygen in mmHg)
Assessment of pulmonary function | 30 days
  Pulmonary function will be assessed by arterial measurement of blood gases (arterial partial pressure of carbon dioxide in mmHg)
Assessment of pulmonary function | 30 days
  Pulmonary function will be assessed by arterial measurement of lactate levels (in mmol/L)
Assessment of hepatic function | 30 days
  Hepatic function will be assessed by laboratory measurements in blood. Changes in aspartate aminotransferase (AST in IU/L) will be measured.
Assessment of hepatic function | 30 days
  Hepatic function will be assessed by laboratory measurements in blood. Changes in alanine aminotransferase (ALT in IU/L) will be measured.
Assessment of hepatic function | 30 days
  Hepatic function will be assessed by laboratory measurements in blood. Changes in gamma-glutamyl transpeptidase (γ-GT in IU/L) will be measured.
Assessment of hepatic function | 30 days
  Hepatic function will be assessed by laboratory measurements in blood. Changes in bilirubin in mg/dL will be measured.
Assessment of hepatic function | 30 days
  Hepatic function will be assessed by laboratory measurements in blood. Changes in fibrinogen in mg/dL will be measured.
Assessment of hepatic function | 30 days
  Hepatic function will be assessed by laboratory measurements in blood. Changes in d-dimers in ng/ml will be measured.
Assessment of renal function | 30 days
  Urine volume during 24 hours (in ml) will be recorded.
Assessment of renal function | 30 days
  Changes in urea (in mg/dL) will be recorded.
Assessment of renal function | 30 days
  Changes in uric acid (in mg/dL) will be recorded.
Assessment of renal function | 30 days
  Changes in creatinine (in mg/dL) will be recorded.
Assessment of cardiac function | 30 days
  Echocardiographic assessment of cardiac left ventricular ejection fraction (LVEF, %)
Assessment of cardiac injury | 30 days
  Measurements of cardiac troponin I (in μg/L) will be used to assess myocardial injury
Assessment of the course of COVID-19 infection | 30 days
  COVID-19 infection will be assessed by inflammatory indices in blood (white blood cells in number per μL)
Assessment of the course of COVID-19 infection | 30 days
  COVID-19 infection will be assessed by inflammatory indices in blood (CRP in mg/L)
Assessment of the course of COVID-19 infection | 30 days
  COVID-19 infection will be assessed by inflammatory indices in blood (erythrocyte sedimentation rate in mm/hr)
Assessment of the course of COVID-19 infection | 30 days
  COVID-19 infection will be assessed by temperature monitoring (in degrees Celsius)
Assessment of the course of COVID-19 infection | 30 days
  COVID-19 infection will be assessed by time needed (in days) for the patient to become negative in COVID-19
Assessment of clinical outcome and safety | 30 days
  Number of participants with major (death, cardiac Arrest, electromechanical dissociation, pulmonary embolism, new myocardial infarction, stroke, pulmonary edema, cardiogenic shock and hypotension, septic shock, pulmonary embolism, serious bleeding) events be recorded during the follow up period
Assessment of clinical outcome and safety | 30 days
  Number of participants with minor (myocarditis, Venous Thromboembolism, left Ventricular mural thrombus, renal failure, hepatic failure, stress ulcers, minor bleeding, paroxysmal supraventricular tachycardia and atrial fibrillation, rhythm disturbances) events will be recorded during the follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Kostopanagiotou, MD, Principal Investigator — ATTIKON University General Hospital
Locations (1):
- Attikon University General Hospital, Haidari/Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pantos C, Apostolaki V, Kokkinos L, Trikas A, Mourouzis I. Acute triiodothyronine treatment and red blood cell sedimentation rate (ESR) in critically ill COVID-19 patients: A novel association? Clin Hemorheol Microcirc. 2021;79(3):485-488. doi: 10.3233/CH-211215. PMID 34151781
- [Derived] Pantos C, Kostopanagiotou G, Armaganidis A, Trikas A, Tseti I, Mourouzis I. Triiodothyronine for the treatment of critically ill patients with COVID-19 infection: A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Jun 26;21(1):573. doi: 10.1186/s13063-020-04474-0. PMID 32586399